CLINICAL TRIAL: NCT01708070
Title: Trial of Asthma Self-Management Education in Patients With Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HL 098240
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Asthma; Depression; Anxiety
Keywords: asthma; depression; anxiety
MeSH Terms: conditions — Asthma; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asthma self-management experimental (Active Comparator): The intervention will involve a self-management workbook, contracting to improve self-management behaviors, instruction in using of a peak flow meter, and follow-up discussions based on the workbook.
  Interventions: Behavioral: Asthma self-management
- Asthma self-management control (Other): The control state will involve a self-management workbook and contracting to improve self-management behaviors.
  Interventions: Behavioral: Asthma self-management

INTERVENTIONS:
Behavioral: Asthma self-management — Patients in the intervention group will receive an asthma workbook, will make a contract to adopt behaviors they think will improve asthma, will be taught how to use a peak flow meter and specific chapters of the workbook will be used as templates for focused instruction during telephone follow-ups which will occur every week for 8 weeks and then approximately every 2 months.

SUMMARY:
Although depressive and anxious symptoms are common in asthma patients and are associated with worse clinical and resource utilization outcomes, there have been no studies focusing on the particular challenges of improving asthma self-management in this population. The investigators hypothesize that a tailored intervention to improve asthma self-management in patients with a known history of depressive and anxious symptoms will be effective in improving asthma-related quality of life.

DETAILED DESCRIPTION:
Depressive and anxious conditions are common during the lifetime of asthma patients and have been shown to be associated with worse asthma as defined by more symptoms, more hospitalizations and greater use of medications. There have been few studies trying to improve asthma outcomes in patients with known depression. One method to improve outcomes is to instruct patients in ways to better self manage asthma. The goal of this study is to test a comprehensive intervention to improve asthma self-management by increasing knowledge and self-efficacy in patients with a known history of a positive screen for depression. Patients will be randomized to two groups - a control group and an intervention group. Patients in the control group will receive an asthma workbook, will make a contract to adopt behaviors they think will improve asthma, and will receive telephone follow-ups approximately every week for 8 weeks and then approximately every 2 months. Patients in the intervention group will receive these components plus they will be taught how to use a peak flow meter and specific chapters of the workbook will be used as templates for focused instruction during telephone follow-ups. The primary outcome will be a comparison of within-patient change in asthma-related quality of life between groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* known history of depressive or anxious symptoms

Exclusion Criteria:

* pregnant
* has cognitive deficits
* no access to telephone

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in asthma-related quality of life | Approximately 12 months
  The primary outcome will be a comparison of within-patient change in Asthma Quality of Life Questionnaire scores between groups.

SECONDARY OUTCOMES:
Number of urgent resource utilization visits for asthma | Approximately 12 months
  An additional outcome will be the comparison of the number or urgent resource utilization visits for asthma.

OTHER OUTCOMES:
Severity of depressive symptoms | Approximately 12 months
  We will characterize and monitor the severity of depressive symptoms during the trial using standardized scales.

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Weill Cornell Internal Medicine Associates/Hospital for Special Surgery, New York, New York, United States